CLINICAL TRIAL: NCT00005266
Title: Cardiovascular Disease Mortality in The NAS-NRC Twin Registry
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1150; R03HL046115 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Diabetes Mellitus; Obesity; Coronary Disease; Myocardial Ischemia
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Diabetes Mellitus; Obesity; Coronary Disease; Myocardial Ischemia

SUMMARY:
To analyze cardiovascular disease mortality and total mortality in the NAS-NRC Twin Registry using a new methodology that allowed for censored observations of outcomes, environmental covariates, and unmeasured genotype-environment interactions.

DETAILED DESCRIPTION:
BACKGROUND:

Methodologically, statistical methods in genetics and epidemiology have developed largely independently; and as a result, there seemed to be little communication between the two fields. Some of the most important hypotheses regarding familial aggregation of chronic diseases related to gene-environment interactions which drew on both fields. The method of analysis used in this study dealt simultaneously with survival time nature of the outcome variable, multiple and continuous environmental risk factors, and correlation in outcomes between related individuals.

The study was supported by the Small Grants Program established by the National Heart, Lung, and Blood Institute in January 1990 to extend analyses of research data generated by clinical trials, population research, and demonstration and education studies.

DESIGN NARRATIVE:

Data available from two epidemiologic questionnaires administered ten years apart were used to determine the extent to which an increased familial risk in cardiovascular disease mortality among twins was mediated by similarities in behavioral risk factors such as smoking, diet, weight changes, physical activity, and socioeconomic variables. The contributions of genetic and environmental factors to twin similarities in health behavior were also examined.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-09; Study Completion 1992-09 (Actual)

REFERENCES:
- [Background] Carmelli D, Swan GE, Robinette D, Fabsitz R. Genetic influence on smoking--a study of male twins. N Engl J Med. 1992 Sep 17;327(12):829-33. doi: 10.1056/NEJM199209173271201. PMID 1508241
- [Background] Carmelli D, Swan GE, Cardon LR. Genetic mediation in the relationship of education to cognitive function in older people. Psychol Aging. 1995 Mar;10(1):48-53. doi: 10.1037//0882-7974.10.1.48. PMID 7779316
- [Background] Swan GE, Carmelli D. Characteristics associated with excessive weight gain after smoking cessation in men. Am J Public Health. 1995 Jan;85(1):73-7. doi: 10.2105/ajph.85.1.73. PMID 7832265
- [Background] Carmelli D, Cardon LR, Fabsitz R. Clustering of hypertension, diabetes, and obesity in adult male twins: same genes or same environments? Am J Hum Genet. 1994 Sep;55(3):566-73. PMID 8079995
- [Background] Carmelli D, Selby JV, Quiroga J, Reed T, Fabsitz RR, Christian JC. 16-year incidence of ischemic heart disease in the NHLBI twin study. A classification of subjects into high- and low-risk groups. Ann Epidemiol. 1994 May;4(3):198-204. doi: 10.1016/1047-2797(94)90097-3. PMID 8055120
- [Background] Carmelli D, Robinette D, Fabsitz R. Concordance, discordance and prevalence of hypertension in World War II male veteran twins. J Hypertens. 1994 Mar;12(3):323-8. PMID 8021487
- [Background] Carmelli D, Swan GE, Robinette D. The relationship between quitting smoking and changes in drinking in World War II veteran twins. J Subst Abuse. 1993;5(2):103-16. doi: 10.1016/0899-3289(93)90055-g. PMID 8400834
- [Background] Carmelli D, Heath AC, Robinette D. Genetic analysis of drinking behavior in World War II veteran twins. Genet Epidemiol. 1993;10(3):201-13. doi: 10.1002/gepi.1370100306. PMID 8349101